CLINICAL TRIAL: NCT00483535
Title: An Open, Repeat Dose Study to Investigate the Effect of Co-administration of the Combined Oral Contraceptive Pill (COC) and GW273225 on the Pharmacokinetics of the COC and to Investigate the Effects of the COC on the Pharmacokinetics of GW273225 in Healthy Female Subjects
Brief Title: Oral Contraceptive Interaction Study for GW273225
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEC107110
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Bipolar Disorder
Keywords: Gw273225, Oral Contraceptive Interaction
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sequence ABC (Experimental): All subjects will receive the treatment sequence ABC where A=combined oral contraceptive pill (COC), B=COC plus GW273225 and C=GW273225. COC will be administered in two cycles that is, cycle 1 (Days 1-21) and cycle 2 (Days 29-49) of the study. The cycles will be separated by a 7 day washout period. GW273225 will be administered at a dose of one 25 milligram tablet once daily on Days 29-75 of the study.
  Interventions: Drug: GW273225; Drug: COC

INTERVENTIONS:
Drug: GW273225 — GW273225 will be available as 25 milligram tablets.
Drug: COC — COC will consist of Microgynon 30 which is available as ethinylestradiol 30 micrograms/levonorgestrel 150 micrograms beige color, sugar-coated tablets.

SUMMARY:
GW273225 is in development for epilepsy and bipolar disorder and can affect women of child bearing potential. A clear understanding of the potential interaction between oral contraceptives and GW273225 is therefore important for clinical investigation of GW273225 in a large number of patients. This study will investigate whether there is any effect of GW273225 upon the components of combined oral contraceptive, and also whether taking oral contraceptives affects the pharmacokinetics (PK) of GW273225.

26 healthy female subjects, aged 18-45 years will take an oral contraceptive (150ug levonorgestrel and 30ug ethinylestrdiol; The study will include a screening period, two cycles on oral contraceptive with GW273225 at 25 mg once per day administered from the start of the second COC cycle for 47 days. There will be a follow-up visit 14-21 days later.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects aged between 18 and 45 years, inclusive.
* Body weight >50 kg and Body Mass Index (BMI) within the range 19-29.9 kg/m2 inclusive.
* Female subjects of child bearing potential will be eligible to participate if they are established on a Microgynon 30 or Ovranette for the previous month
* If taking a similar ethinyl oestradiol dose (30 or 35 mcg) combined with a progestogen at fixed dose for 21 days then willing to switch to Microgynon 30
* Subjects will use additional contraception as described in the protocol. One of the methods listed in the protocol is acceptable in conjunction with COC as the method of contraception if there is indisputable data that it is >99% effective, otherwise it should be used with a barrier method (condom or occlusive cap (diaphragm or cervical/vault caps) used with spermicidal foam/gel/film/cream/suppository).
* Subjects must smoke ≤ 10 cigarettes per day.
* No abnormality on relevant clinical examination. A subject with a clinical abnormality may be included only if the Investigator in consultation with the GSK Medical Monitor considers that the abnormality will not introduce additional risk factors and will not interfere with the study procedures.
* No abnormality on relevant clinical chemistry or haematology examination at the pre-study medical examination. Subjects with laboratory parameters outside the reference range for this age group will only be included if the Investigator in consultation with the GSK Medical Monitor considers that such findings will not introduce additional risk factors.
* A 12-lead ECG and vital signs at the pre-study medical examination, which are normal. (including QTc which is <450msec)
* The subject has signed and dated written informed consent prior to admission to the study
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

* History or evidence of drug or alcohol abuse within six months of study start.
* Weekly alcohol intake of more than 14 units or an average daily intake of greater than 2 units.
* Female subject pregnant (positive serum human chorionic gonadotrophin (hCG) test at screening) or lactating. HIV, Chronic hepatitis B and C, as evidenced by positive Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody
* Subject has received prescribed or non-prescribed medication (including vitamins and herbal remedies) within 14 days prior to day 1 which in the opinion of the investigator, could have interfered with the study procedures or compromised safety.
* History of gastro-intestinal, hepatic or renal disease or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* History of thrombotic events or presence of significant risk factors for thrombosis.
* Supine Blood Pressure greater than or equal to 140/90.
* Progestogen- releasing IUD contraceptive.
* Participation in a trial with any drug within 84 days before the start of the study.
* Donation of more than 1500 mL blood in the previous 12 months.
* History or presence of any condition contra-indicated to combined oral contraceptive.
* Any subject where the potential side effects of GW273225 could affect their professional occupation, e.g. operating machinery, driving.
* Any subjects who cannot refrain from driving for the duration of administration of GW273225 and for 3 days afterwards.
* History of clinically relevant skin rashes that, in the opinion of the investigator, might interfere with the conduct of the study.
* Subject has current or past history of seizure disorder or brain injury (traumatic or disease-related), or any condition which, in the opinion of the investigator, predisposes to seizure; subject treated with other medications or treatment regimens that lower seizure threshold; subject undergoing abrupt discontinuation of alcohol or sedatives (including benzodiazepines).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-03-07 (Actual); Primary Completion 2007-11-16 (Actual); Study Completion 2007-11-16 (Actual)

PRIMARY OUTCOMES:
0-24hrs PK of oral contraceptive components | 0-24hrs

SECONDARY OUTCOMES:
0-24hrs PK of GW273225 Hormone levels with co-administration of oral contraceptive and GW273225 | 0-24hrs
blood drug levels of GW273225 in the presence or absence of the Combined Oral Contraceptive (COC) | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours post dosing on Day 49 and Day 75
blood levels of ethinylestradiol and levonorgestrel of the COC in the presence or absence of GW273225. | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours post dosing on Day 21 and Day 49
blood levels of FSH, LH and progesterone | Up to Day 45
blood levels of Oestradiol and SBHG | Up to Day 45
Electrocardiogram (ECG) recordings | Up to Day 96
Adverse events | Up to Day 96
Vital signs | Up to Day 96

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- See also: Results for study 107110 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/NEC107110?search=study&search_terms=107110#rs